CLINICAL TRIAL: NCT02327481
Title: Randomized Controlled Trials Comparing Clinical Outcomes of 3D Versus 2D Laparoscopic Surgery for Gastric Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fujian Medical University (Other)
Responsible Party: Principal Investigator, Chang-Ming Huang, Prof., Fujian Medical University Union Hospital, Fujian Medical University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: FUGES-001
Record Dates: First submitted 2014-12-24; First posted 2014-12-30 (Estimated); Last update posted 2023-04-07 (Actual); Status verified 2023-04

CONDITIONS: Stomach Neoplasms
Keywords: Stomach Neoplasms Laparoscopy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 3D Laparoscopic Surgery (Experimental): 3D Laparoscopic Surgery will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: 3D Laparoscopic Surgery
- 2D Laparoscopic Surgery (Active Comparator): 2D Laparoscopic Surgery will be performed for the treatment of patients assigned to this group.
  Interventions: Procedure: 2D Laparoscopic Surgery

INTERVENTIONS:
Procedure: 3D Laparoscopic Surgery — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, 3D laparoscopic gastrectomy will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience.
  Arms: 3D Laparoscopic Surgery
Procedure: 2D Laparoscopic Surgery — After exclusion of T4b, bulky lymph nodes, or distant metastasis case by diagnostic laparoscopy, 2D laparoscopic gastrectomy will be performed with curative treated intent. The type of reconstruction will be selected according to the surgeon's experience.
  Arms: 2D Laparoscopic Surgery

SUMMARY:
The purpose of this study is to explore the feasibility, safety, and efficacy of 3D Laparoscopic Surgery for Gastric Cancer. The patients with gastric adenocarcinoma (cT1-4aN0-3M0) were studied.

DETAILED DESCRIPTION:
A prospective randomized comparison of 3D and 2D laparoscopic surgery for gastric cancer will be performed, to evaluate the clinical value and provide theoretical basis and clinical experience for the extensive application of the 3D laparoscopic technique. The evaluation parameters are perioperative clinical efficacy, postoperative life quality, immune function and 3-year/5-year survival and recurrence rates.

ELIGIBILITY:
Inclusion Criteria:

* (1)Age from over 19 to under 74 years
* (2)cT1-4a(clinical stage tumor), N0-3, M0 at preoperative evaluation according to the American Joint Committee on Cancer (AJCC) Cancer Staging Manual Seventh Edition
* (3)Heart, lungs, kidneys, and other vital organs function well, with no obvious surgical contraindications
* (4)Preoperative examination with no distant metastasis, no significantly enlarged lymph nodes around the main abdominal artery, and tumor not a direct violation of the pancreas, spleen, and other surrounding organs
* (5)American Society of Anesthesiology (ASA) score class I, II, or III
* (6)Written informed consent

Exclusion Criteria:

* (1)Women during pregnancy or breast-feeding
* (2)Severe mental disorder
* (3)History of previous upper abdominal surgery (except laparoscopic cholecystectomy)
* (4)Enlarged splenic hilar lymph nodes with integration into a mass and surrounding the blood vessels
* (5)History of unstable angina or myocardial infarction within the past six months
* (6)History of cerebrovascular accident within the past six months
* (7)History of continuous systematic administration of corticosteroids within one month
* (8)History of previous neoadjuvant chemotherapy or radiotherapy
* (9)T4b tumors
* (10)Emergency surgery due to complication (bleeding, obstruction, or perforation) caused by gastric cancer
* (11)FEV1(Forced expiratory volume in one second)<50% of predicted values

Ages: 19 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 438 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2016-04-26 (Actual); Study Completion 2021-04-26 (Actual)

PRIMARY OUTCOMES:
Operating time | 1 day
  Operating time

SECONDARY OUTCOMES:
Intraoperative situation | 1 day
  The number of lymph node dissection, the number of positive lymph nodes, intraoperative lymph node dissection time(regional analysis: infrapyloric area lymph node, suprapancreatic area lymph node, splenic hilar area lymph node, cardial area lymph node), intracavitary anastomosis time(patients who undergo totally laparoscopic surgery are analyzed), intraoperative blood loss, intraoperative injury, the amount of use of titanium clip, the rate of conversion to laparotomy
Postoperative recovery course | 10 days
  Time to first ambulation, flatus, liquid diet and soft diet, duration of postoperative hospital stay and postoperative pain are used to assess the postoperative recovery course.Visual analog pain score method is used to evaluate the difference of postoperative pain degree.
Complication | 30 days;36 months
  Early complications occurred within 30 days after operation: pulmonary infection, incision complication, intestinal obstruction, abdominal infection, anastomotic bleeding, anastomotic fistula, gastric emptying; Long-term complications (30 days later after operation): anastomotic stenosis, intestinal obstruction, dumping syndrome
The postoperative pathology | 7 days
  The postoperative pathological type and pTNM stage.
Inflammatory and immune response | 7 days
  The daily highest body temperature before discharge and the values of white blood cell count, hemoglobin, C-reactive protein, prealbumin and relevant immune cytokines including T cell percentage, T-helper lymphocytes (CD4+) percentage, T-suppressor lymphocytes (CD8+) percentage, natural killer (NK) cells percentage from peripheral blood before operation and on postoperative day 1, 3, 5 are recorded.
Morbidity and mortality | 30 days;36 months
  The early postoperative complication and mortality are defined as the event observed within 30 days after surgery, while the time frame for late complication is the period from postoperative day 31th to the end of month 36th.
Hospitalization expenses | 1 months
  The cost from admission to discharge
3-year disease free survival rate | 36 months
  Disease-free survival was defined as the time from surgery to the time of recurrence or death from any cause
3-year overall survival rate | 36 months
  Overall survival was defined as the time from surgery to death from any cause
5-year disease free survival rate | 60 months
  Disease-free survival was defined as the time from surgery to the time of recurrence or death from any cause
5-year overall survival rate | 60 months
  Overall survival was defined as the time from surgery to death from any cause
Recurrence patterns | 60 months
  Recurrence patterns are classified into five categories at the time of first diagnosis: locoregional, hematogenous, peritoneal, distant lymph node, and mixed type.

CONTACTS AND LOCATIONS:
Overall Officials: Changming Huang, M.D.,Ph.D., Study Chair — Fujian Medical University Union Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Wei LH, Zheng HL, Liu ZY, Du XQ, Chen CS, Xu BB, Zheng HH, Lin GT, Xie JW, Zheng CH, Wang JB, Huang CM, Li P. Preoperative visceral fat area predicts intraoperative adverse events during lymphadenectomy in laparoscopic gastrectomy for gastric cancer: a post hoc analysis. Surg Endosc. 2025 Apr;39(4):2275-2287. doi: 10.1007/s00464-025-11602-x. Epub 2025 Feb 12. PMID 39937241
- [Derived] Xu BB, Zheng HL, Chen CS, Xu LL, Xue Z, Wei LH, Zheng HH, Shen LL, Zheng CH, Li P, Xie JW, Lin JX, Zheng YH, Huang CM. Development and validation of a preoperative radiomics-based nomogram to identify patients who can benefit from splenic hilar lymphadenectomy: a pooled analysis of three prospective trials. Int J Surg. 2024 Jul 1;110(7):4053-4061. doi: 10.1097/JS9.0000000000001337. PMID 38980664
- [Derived] Zhong Q, Chen JY, Shang-Guan ZX, Liu ZY, Lin GT, Wu D, Jiang YM, Wang JB, Lin JX, Chen QY, Lin JL, Xie JW, Li P, Lu J, Huang CM, Zheng CH. Long-term oncological outcomes of 3D versus 2D laparoscopic gastrectomy for gastric cancer: a randomized clinical trial. Gastric Cancer. 2024 May;27(3):598-610. doi: 10.1007/s10120-024-01470-0. Epub 2024 Feb 20. PMID 38379100
- [Derived] Liu ZY, Chen QY, Zhong Q, Li P, Xie JW, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Huang CM, Zheng CH. Intraoperative Adverse Events, Technical Performance, and Surgical Outcomes in Laparoscopic Radical Surgery for Gastric Cancer: A Pooled Analysis From 2 Randomized Trials. Ann Surg. 2023 Aug 1;278(2):222-229. doi: 10.1097/SLA.0000000000005727. Epub 2022 Oct 17. PMID 36250322
- [Derived] Lu J, Xu Y, Wu Y, Huang XY, Xie JW, Wang JB, Lin JX, Li P, Zheng CH, Huang AM, Huang CM. Tumor-infiltrating CD8+ T cells combined with tumor-associated CD68+ macrophages predict postoperative prognosis and adjuvant chemotherapy benefit in resected gastric cancer. BMC Cancer. 2019 Sep 14;19(1):920. doi: 10.1186/s12885-019-6089-z. PMID 31521128
- [Derived] Liu ZY, Chen QY, Zhong Q, Xie JW, Wang JB, Lin JX, Lu J, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Zheng HL, Zheng CH, Huang CM, Li P. Is three-dimensional laparoscopic spleen preserving splenic hilar lymphadenectomy for gastric cancer better than that of two-dimensional? Analysis of a prospective clinical research study. Surg Endosc. 2019 Oct;33(10):3425-3435. doi: 10.1007/s00464-018-06640-7. Epub 2019 Feb 26. PMID 30809728
- [Derived] Xu BB, Lu J, Zheng ZF, Xie JW, Wang JB, Lin JX, Chen QY, Cao LL, Lin M, Tu RH, Huang ZN, Lin JL, Zheng CH, Huang CM, Li P. The predictive value of the preoperative C-reactive protein-albumin ratio for early recurrence and chemotherapy benefit in patients with gastric cancer after radical gastrectomy: using randomized phase III trial data. Gastric Cancer. 2019 Sep;22(5):1016-1028. doi: 10.1007/s10120-019-00936-w. Epub 2019 Feb 9. PMID 30739259
- [Derived] Zheng CH, Lu J, Zheng HL, Li P, Xie JW, Wang JB, Lin JX, Chen QY, Cao LL, Lin M, Tu RH, Huang CM. Comparison of 3D laparoscopic gastrectomy with a 2D procedure for gastric cancer: A phase 3 randomized controlled trial. Surgery. 2018 Feb;163(2):300-304. doi: 10.1016/j.surg.2017.09.053. Epub 2017 Nov 28. PMID 29195739
- [Derived] Lu J, Zheng CH, Zheng HL, Li P, Xie JW, Wang JB, Lin JX, Chen QY, Cao LL, Lin M, Tu RH, Huang CM. Randomized, controlled trial comparing clinical outcomes of 3D and 2D laparoscopic surgery for gastric cancer: an interim report. Surg Endosc. 2017 Jul;31(7):2939-2945. doi: 10.1007/s00464-016-5310-2. Epub 2016 Nov 8. PMID 27826781